CLINICAL TRIAL: NCT02805491
Title: Case-control Study of the Influence of Pesticide Exposure on the Occurrence of Hypospadias in Newborns in Picardie
Brief Title: Influence of Pesticide Exposure on the Occurrence of Hypospadias in Newborns in Picardie
Acronym: HYPOMECO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI10-DR-HARAUX
Record Dates: First submitted 2016-06-08; First posted 2016-06-20 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Hypospadias
Keywords: Hypospadias; newborns; pesticide; Picardie
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — meconium
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with hypospadias: parent-child triads as cases (male newborns with hypospadias)
  Interventions: Other: meconium; Other: self questionnaires to parents
- without hypospadias: parent-child triads as controls (male newborns without hypospadias)
  Interventions: Other: meconium; Other: self questionnaires to parents

INTERVENTIONS:
Other: meconium — to evaluate internal exposure to pesticide
Other: self questionnaires to parents — to evaluate external exposure to pesticide

SUMMARY:
We want to see if there is a relationship between exposure to pesticides and the occurrence of hypospade in Picard newborn .

DETAILED DESCRIPTION:
Hypospadias is the most frequent malformation of the external genital organs in the male infant. Incomplete virilization of the genital bud results in hypoplasia of the tissues on the ventral aspect of the penis, with an ectopic ureteral meatus, a curved penile shaft and an incompletely formed foreskin. The condition is generally isolated and the aetiology is unknown. The pathogenesis is complex and involves hormonal, genetic and environmental factors (which are probably interlinked).

A doubling in the incidence of hypospadias over the last 15 years has emphasized the probable role of environment factors: in fact, certain exogenous compounds (collectively referred to as "endocrine disruptors" (EDs)) may modify hormonal functions and thus exert harmful effects on the organism or its offspring.

The male urethra develops between the 8th and 16th weeks of gestation in an androgen-dependence manner. In utero exposure of the foetus to EDs may have a physiopathological role in the abnormal development of the male genital bud and thus in the development of hypospadia. These EDs are present in many different substances, such as pesticides.

Many epidemiological studies have evidenced an increase in the incidence of hypospadias in children born to exposed parents. Furthermore, animal studies have identified a certain number of compounds associated with hypospadias after in utero exposure. However, human foetal samples have very rarely been assayed in an attempt to measure the true level of impregnation (i.e. the dose received). At present, it is not possible to draw firm conclusions with regard to the true extent of a link between EDs and the increased incidence of hypospadia.

The "HypoMeco" project is a prospective case-control study.

ELIGIBILITY:
Inclusion Criteria:

* male newborns
* born after February 1st, 2011, in a maternity hospital/clinic in the Picardie region

Exclusion Criteria:

* refusal to participate,
* severe associated disorders
* associated multiple malformation syndromes
* patients not attending the consultation.
* parents under the age of 18
* prison inmates

Ages: 1 Minute to 1 Day | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: parent-child triads as cases (male newborns with hypospadias) and parent-child triads as controls (male newborns without hypospadias)
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2014-12-20 (Actual); Study Completion 2014-12-20 (Actual)

PRIMARY OUTCOMES:
presence of hypospadia | 1 month
  to compare the incidence of hypospadias in newborns in the Picardie region exposed to pesticides and in those not exposed.

SECONDARY OUTCOMES:
prevalence of hypospadias and each of its forms in the Picardie region | 1 year
  meconium analysis
the proportions of associated endocrine disorders (regardless of the severity of hypospadias) through systematic screening. | 1 year
  meconium analysis
levels of endocrine disruptors | day 1 , 1 month
  meconium analysis

CONTACTS AND LOCATIONS:
Overall Officials: Elodie HARAUX, PhD, Principal Investigator — CHU Amiens
Locations (11):
- France (11):
  - CH Abbeville, Abbeville
  - CHU Amiens, Amiens
  - Groupe Santé Victor Pauchet, Amiens
  - CH Chauny, Chauny
  - CH Chateau Thierry, Château-Thierry
  - CH Compiegne, Compiègne
  - CH Creil, Creil
  - CH Laon, Laon
  - CH Péronne, Péronne
  - CH Saint Quentin, Saint-Quentin
  - CH Senlis, Senlis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haraux E, Tourneux P, Kouakam C, Stephan-Blanchard E, Boudailliez B, Leke A, Klein C, Chardon K. Isolated hypospadias: The impact of prenatal exposure to pesticides, as determined by meconium analysis. Environ Int. 2018 Oct;119:20-25. doi: 10.1016/j.envint.2018.06.002. Epub 2018 Jun 18. PMID 29929047